CLINICAL TRIAL: NCT03170323
Title: A Prospective Randomized, Controlled Trial of Mycophenolate Mofetil Plus Steroid in the Treatment Of Patients With Progressive Idiopathic Membranous Nephropathy
Brief Title: Mycophenolate Mofetil Plus Steroid in the Treatment Of Patients With Progressive Idiopathic Membranous Nephropathy
Acronym: MMF-STOP-IMN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GGH2016430H
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-02

CONDITIONS: Idiopathic Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Mycophenolic Acid; Cyclosporins

STUDY DESIGN:
Intervention Model Description: Drug: Mycophenolate mofetil, high dose steroid Drug: Cyclosporin, low dose steroid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mycophenolate mofetil (Experimental): Drug: Mycophenolate mofetil, high dose steroid Duration: 1 year
  Interventions: Drug: Mycophenolate Mofetil
- Cyclosporin (Active Comparator): Drug: Cyclosporin, low dose steroid Duration: 1 year
  Interventions: Drug: Cyclosporins

INTERVENTIONS:
Drug: Mycophenolate Mofetil — steroid 1mg/kg/d and Mycophenolate mofetil 500mg bid
  Arms: Mycophenolate mofetil
Drug: Cyclosporins — steroid 0.15mg/kg/d and Cyclosporin 3-5mg/kg/d
  Arms: Cyclosporin

SUMMARY:
Idiopathic membranous nephropathy (IMN) remains a common cause of the nephrotic syndrome in adults. There are few randomized clinical trials regarding the therapeutic effect of mycophenolate mofetil in patients with Idiopathic membranous nephropathy. This study aims to evaluate whether treatment with mycophenolate mofetil is non-inferior to cyclosporins in inducing long-term remission (complete or partial) of proteinuria in patients with idiopathic membranous nephropathy.

DETAILED DESCRIPTION:
Idiopathic membranous nephropathy is the most common cause of nephrotic syndrome in adults. In recent year, IMN remains one of the most common glomerular diseases. Long-term remission and stable renal function can prevent idiopathic membranous nephropathy from progressing to end-stage renal disease. Cyclosporine and cyclophosphamide are recommended to be first-line treatment regimen. Corticosteroid is the basic combined drug in the treatment of idiopathic membranous nephropathy. Mycophenolate mofetil is a recently developed immunosuppressive agent with fewer renal toxicity than cyclosporin.Besides, high dose prednisone may be effective for patients in Asia according to literatures from Asia. In our study, patients with idiopathic membranous nephropathy would be treated with mycophenolate mofetil and high dose prednisone,whose outcome will be compared with cyclosporin and low dose prednisone. We aims to evaluate whether treatment with mycophenolate mofetil is non-inferior to cyclosporins in inducing long-term remission of proteinuria in patients with idiopathic membranous nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients who provided informed consent
* 2.Patients who are diagnosed as membranous nephropathy by renal biopsy,and other secondary factors are excluded
* 3.18 years of age or older, male or female
* 4.24 hours urine protein or spot urine protein/creatinine ratio > 8.0 g/day at least for twice confirmed
* 5.The patients that satisfy more than three of following items are included even if proteinuria is less than 8 grams per day:

  1. estimated glomerular filtration rate(eGFR) < 60 ml/min/1.73m2
  2. Hypertension (BP above 140/90millimetre of mercury or BP above 120/80millimetre of mercury in patients taking anti-hypertensive agents)
  3. 24 hours urine protein or spot urine protein/creatinine ratio > 5.0 g/day
  4. Serum albumin (g/dL) < 3.0

Exclusion Criteria:

* 1.Severe infective disease
* 2.Allergy history to clinical trial medication and acute or chronic allergy for 4 weeks recently.
* 3.Clinical history of treatment with other immunosuppressive medication
* 4.Probability of pregnancy, breast feeding woman
* 5.Uncontrolled hypertension (more than 160/100 millimetre of mercury )
* 6.estimated glomerular filtration rate(eGFR)<30 ml/min/1.73m2。
* 7.Abnormal liver function test (more than 3 times above compared with normal value)
* 8.Absolute neutrophil count <1,500/mm3 or leukocyte <2,500/mm3 or platelets <100,000/mm3
* 9.Secondary membranous nephropathy
* 10.Expected life expectancy is less than 1 year
* 11.The researchers evaluated that the patient's compliance was not appropriate for the trial
* 12.Previous or present history of cancer and have risk of recurrence or metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Remission | after treatment for 1 year.
  Urinary protein excretion<0.3 g/d (uPCR<300 mg/g or <30 mg/mmol), confirmed by two values at least 1 week apart, accompanied by a normal serum albumin concentration, and a normal serum creatinine.
Partial Remission | after treatment for 1 year.
  Urinary protein excretion <3.5 g/d (uPCR <3500 mg/g or <350 mg/mmol) and a 50% or greater reduction from peak values;confirmed by two values at least 1 week apart, accompanied by an improvement or normalization of the serum albumin concentration and stable serum creatinine.

SECONDARY OUTCOMES:
estimated Glomerular Filtration Rate | after treatment for 1 year
  time to a 50% reduction in baseline estimated Glomerular Filtration Rate (according to CKD-EPI)
serum creatinine | after treatment for 1 year
  time to doubling of baseline creatinine

CONTACTS AND LOCATIONS:
Overall Officials: xinling Liang, M.D.,PH.D, Principal Investigator — Nephrology Dept,Guangdong General Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952